CLINICAL TRIAL: NCT03922243
Title: Dental Treatments Analysis Rendered by Undergraduates at Ajman University, Fujairah, Uae
Brief Title: An Analysis of Dental Treatments Rendered by Undergraduates at Ajman University to Patients From Fujairah, Uae
Status: Completed | Type: Observational
Sponsor: Ajman University (Other)
Responsible Party: Principal Investigator, suleiman omar ergieg, Professor, Ajman University
Other Study IDs: 2017-FJ-DN-03
Record Dates: First submitted 2019-03-17; First posted 2019-04-19 (Actual); Last update posted 2019-04-19 (Actual); Status verified 2019-04

CONDITIONS: Treatment
Keywords: students; dental treatment; gender; age
MeSH Terms: conditions — Coitus | interventions — Retrospective Studies

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: retrospective — Retrospective study to assess treatment done by dental students

SUMMARY:
A total of 650 dental records were selected from 6000 dental records of patients who had received dental treatment in the Dental Clinic, College of Dentistry, Ajman University(AU)-Fujairah Campus, between academic year,2015/2016 and 2016/2017

DETAILED DESCRIPTION:
A total of 650 dental records was randomly selected from 6000 dental records of patients who had received dental treatment in the Dental Clinic, College of Dentistry, Ajman Universi-ty(AU),Fujairah Campus, between the academic years 2015/2016 and 2016/2017. The size of study sample was determined using, Cochran' formula at 95% confidence. Using the random table generated by Microsoft Excel, the records for 650 patients were then randomly selected. After all the dental records to be included in this study were chosen and retrieved from the achieves. The following types of dental treatments: Composite restorations, amalgam restorations, glass ionomer restorations, fixed prosthetic treatments, removable prosthetic treatment, endodontic treatments, extractions treatments, fluoride treatments, fissure sealants treatment, pulp therapy treatments and stainless steel crowns treatments were extracted from the patient's dental records, coded and recorded in Microsoft excel sheet.

ELIGIBILITY:
Inclusion Criteria:

* Dental treatment performed in the time frame

Exclusion Criteria:

* Dental treatment not performed

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: patients registered at Ajman University,Dental clinic,Fujairah
Sampling Method: Non-Probability Sample
Enrollment: 650 (Actual)
Dates: Start 2018-08-10 (Actual); Primary Completion 2019-02-10 (Actual); Study Completion 2019-02-10 (Actual)

PRIMARY OUTCOMES:
Incidences of student performed dental treatment | From baseline to 12 months
  Previous Dental case records used as measurement

CONTACTS AND LOCATIONS:
Locations (1):
- Ajman university, Fujairah, UAE, United Arab Emirates

IPD SHARING:
Plan to Share IPD: Undecided